CLINICAL TRIAL: NCT00822146
Title: Cardiac Resynchronization Therapy (CRT) Efficacy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CEN_G_CA_11
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure
Keywords: CRT
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Device: CRT

INTERVENTIONS:
Device: CRT — classified

SUMMARY:
The aim of this research study is the invasive evaluation of CR therapy efficacy in patients treated with an InSync Sentry device using an external monitoring device to obtain important cardiac parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patient indicated for InSync Sentry CRT device implant
* The patient must be willing and capable of following the study protocol
* EF ≤ 40%
* Systolic pulmonary artery pressure derived by echocardiography > 40
* Patients with their device functioning in a bi-ventricular mode, with defibrillation detection and therapy enabled
* Marked released transvenous RVCoil lead

Exclusion Criteria:

* Patients with chronic AF
* Patients with unipolar atrial or unipolar right ventricular leads
* Patients needing a Lower Rate faster than 110 beats per minute
* Patients with an implanted Medtronic Sentry in whom missing one day's fluid-measurement value is undesirable
* Patients who cannot tolerate turning off Rate Response during the study
* Patients with acute ischemia
* Patients whose InSync Sentry battery is at ERI or EOL status
* Patients with "RAMware" downloaded from other studies
* Patients with medical conditions that would limit study participation
* Patients who are pregnant
* Patients enrolled in another study, which could influence the result of this study
* Patients on the heart transplantation list or patients with transplanted hearts
* Patients is not available for follow-up care
* Patients has not signed a consent form
* Patients with renal failure needing dialysis
* Patients whose compliance can expected to be poor
* Patients with a mechanical tricuspid valve
* Life expectation < 12 months
* Severe PAOD (peripheral arterial occlusive disease)
* Underage patients, pregnant or breast feeding women and female patients not using adequate contraception are excluded from participating in the study

Since right after implantation study procedure will follow, patient has to sign the informed consent before the implantation. However the following criteria are device based and can therefore not checked at time of sign off.

Therefore lead performance will be checked right after the implant and before the study specific procedure. If exclusion criteria are fulfilled patient exit the study and no study specific procedure will be done.

* Patients with non-intact or unstable leads, as indicated on the "Quick Look" screen of the Medtronic Model 2090 programmer by the presence of lead warnings such as the following:

  * LV pacing lead impedance is > 2500 ohms
  * LV pacing lead impedance is < 200 ohms
  * A. pacing lead impedance is > 2500 ohms
  * A. pacing lead impedance is < 200 ohms
  * SVC defib lead impedance is > 200 ohms
  * SVC defib lead impedance is < 20 ohms
  * RV pacing lead impedance is > 2500 ohms
  * RV pacing lead impedance is < 200 ohms
* Patients with atrial pacing thresholds lower than 1.0 volts at .03 ms
* Patients with right ventricular pacing thresholds lower than 1.0 volts at .03 ms
* Patients with left ventricular pacing thresholds lower than 1.0 volts at .03 ms
* Patients in whom a Lower Rate cannot be programmed to achieve consistent atrial pacing for the duration of download software installed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-12; Primary Completion 2011-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
classified | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany